CLINICAL TRIAL: NCT05312892
Title: Sympathetic Mechanisms in the Cardiovascular and Metabolic Alterations of Obesity, Crossover Design Study.
Brief Title: Sympathetic Mechanisms in Obesity-Crossover Design
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 212413
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — Amlodipine; Antihypertensive Agents; moxonidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will received 2 weeks of capsules containing placebo.
  Interventions: Drug: Placebo
- Amlodipine (Active Comparator): Subjects will received 2 weeks of capsules containing amlodipine.
  Interventions: Drug: Amlodipine
- Moxonidine (Experimental): Subjects will received 2 weeks of capsules containing moxonidine.
  Interventions: Drug: Moxonidine

INTERVENTIONS:
Drug: Amlodipine — Subjects will receive either an antihypertensive (amlodipine or moxonidine) medication or placebo for two weeks, then cross over to the second arm, and then after 2 weeks of the second drug/placebo, will be switched to the third arm.
  Other Names: Antihypertensive
  Arms: Amlodipine
Drug: Moxonidine — Moxonidine
  Other Names: Antihypertensive
  Arms: Moxonidine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
We will study obese hypertensive subjects in a randomized, crossover study to determine if two weeks sympathetic blockade improves endogenous glucose production. Subjects will be studied on 3 different occasions after two weeks of receiving either placebo, amlodipine (vasodilator arm) or moxonidine (study arm). The order of the studies will be determined using computer-generated randomization. Patients will be blinded as to which treatment they are receiving on each day. An investigator blinded to the treatment assignment will perform the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races between 18 and 65 years of age
* Hypertension defined by two or more properly measured seated blood pressure readings >130/85 mmHg or currently on antihypertensive medication.
* Obesity will be defined as having a body mass index (BMI) ≥ 30 kg/m2.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy or breast feeding
* Current smokers or history of heavy smoking (>2 packs/day)
* History of alcohol or drug abuse
* Previous allergic reaction to study medications
* Type I diabetes.
* Cardiovascular disease other than hypertension such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy
* History of serious cerebrovascular disease such as cerebral hemorrhage, stroke, or transient ischemic attack
* History or presence of immunological or hematological disorders
* Impaired renal function
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
* Treatment with any investigational drug in the 1 month preceding the study
* Inability to give, or withdraw, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol (i.e., clinically significant abnormalities on clinical, mental examination or laboratory testing or inability to comply with protocol, inability to find IV access)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Endogenous glucose production | During two-step insulin clamp (six hours)
  Rate of appearance and disappearance of labeled glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided